CLINICAL TRIAL: NCT03300492
Title: A Phase I/II Single Center Study to Assess the Safety, Tolerability and Feasibility of Pre-emptive Immunotherapy With in Vitro Expanded Natural Killer Cells in Patients Treated With Haplo-HSCT for AML/MDS
Brief Title: Expanded Natural Killer Cells Following Haploidentical HSCT for AML/MDS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Haplo-NK-DLI for AML/MDS
Record Dates: First submitted 2017-07-30; First posted 2017-10-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Natural Killer cells; NK cells; Immunotherapy; haploidentical hematopoietic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective, single center, open-label, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK-DLI (Experimental): Preemptive immunotherapy with ex vivo expanded NK cells on days
  +10, +15 and +20 with increasing NK cell doses following haplo-HSCT.
  Interventions: Other: NK-DLI

INTERVENTIONS:
Other: NK-DLI — Application of three infusions of ex vivo expanded NK cells on days
  +10, +15 and +20 with increasing NK cell doses (1x107/kg, 1x108/kg and the remaining cells up to 1x109/kg) following haplo-HSCT. Maximal cumulative T-cell dose is fixed at <1x105/kg.

SUMMARY:
The study examines the application of expanded natural killer cells (NK cells) following haploidentical allogeneic hematopoietic stem cell transplantation (haplo-HSCT) for AML or MDS. Haplo-HSCT is a preferred treatment option for patients with AML or MDS without a HLA-matched donor. With administration of cyclophosphamide post-transplant , the safety of the procedure is similar to a HSCT from a HLA-identical donor. Relapse of AML/MDS represents a serious problem following haplo-HSCT. NK cells are immune cells able to destroy tumor cells. Their potency has been established particularly in the setting of a haplo-HSCT. In the current study, study participants undergoing haplo-HSCT will receive expanded NK cells from their respective stem-cell donors following haplo-HSCT. The primary goal of the study is to establish the safety and feasibility of this approach. In addition, the activity of the NK cells will be examined.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* >18 years of age
* No HLA-matched related or unrelated donor available
* AML or MDS-EB with indication for a haplo-HSCT according to the guidelines of the University Hospital Basel Stem Cell Transplant Team
* Judged by the transplant physicians to have adequate organ function and no contraindications to haplo-HSCT
* Available related haploidentical donor
* Written informed consent

Donor:

* >18 years old, haploidentical parent, sibling or other relative
* Donor suitable for cell donation and apheresis according to standard criteria
* Written informed consent

Exclusion Criteria:

Patient:

* APL diagnosis
* Presence of relevant (mean fluorescence intensity >2000) donor-specific anti-HLA antibodies
* Pregnancy
* Necessity of immunosuppression apart from GvHD prophylaxis

Exclusion Criteria:

Donor:

• Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events including GvHD and infections. | 1 year following haplo HSCT
  As defined by the CTCAE version 4.03 and the NIH Scoring of GvHD.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year following haplo HSCT
Incidence of AML/MDS-EB complete morphological and molecular remission (CR) at day + 30, + 90, +180 and 1 year post allo-HSCT | 1 year following haplo HSCT
  rejection.
Incidence of graft rejection | 1 year following haplo HSCT
Number of NK cells given per kg body weight | 30 days following haplo-HSCT
Number of NK-DLI infusions applied | 30 days following haplo-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Passweg, Prof. MD, Principal Investigator — University Hospital Basel, Basel Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No